CLINICAL TRIAL: NCT03300687
Title: First in Human Safety Study of FX-322 in Adults Undergoing Cochlear Implantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Frequency Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: FX-322-103
Record Dates: First submitted 2017-09-15; First posted 2017-10-03 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Subjects will receive FX-322 as an intratympanic injection
  Interventions: Drug: FX-322
- Placebo (Placebo Comparator): Subjects will receive Placebo as an intratympanic injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FX-322 — intratympanic injection
  Arms: Active
Drug: Placebo — intratympanic injection
  Arms: Placebo

SUMMARY:
This is a phase 1 safety study performed in male or female adult participants with an established diagnosis of severe to profound sensorineural hearing loss that meets the criteria for cochlear implantation and the participant has already chosen to undergo cochlear implant surgery.

DETAILED DESCRIPTION:
Approximately 12 participants will be enrolled in the study. Assessed will be safety and tolerability of FX-322 administered by intratympanic injection. Also assessed will be the FX-322 concentration in cochlear fluid (perilymph), the pharmacokinetic (PK) profile of FX-322 to determine the systemic exposure to FX-322.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects with an established diagnosis of severe to profound sensorineural hearing loss audiometric threshold of 80 dB HL or poorer at 500 Hz that meets the criteria for cochlear implantation and the subject has already chosen to undergo cochlear implant surgery.
2. Willingness and ability to comply with scheduled visits, ear examination, drug administration plan, auditory and laboratory tests, study restrictions, and all study procedures.

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

1. Persistent perforation of tympanic membrane or other tympanic membrane disorder that would interfere with the delivery and safety assessment of an intra -tympanic medication or reasonably be suspected to affect tympanic membrane healing after injection.
2. Any conductive component defined as air-bone gaps >10 dB at two or more frequencies.

Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety and Tolerability) of FX-322. | Treatment-emergent adverse events will be assessed over a several hour to two week period
  To assess the incidence of adverse safety events (vertigo, tinnitus, perforation) including severe adverse events.

SECONDARY OUTCOMES:
Plasma Pharmacokinetics | Systemic exposure will be evaluated over a 72 hour period
  Drug exposure in the systemic circulation by evaluating Cmax and AUC Drug exposure evaluated by area under the plasma concentration versus time curve (AUC)
Plasma Pharmacokinetics | Within a 24 hour period after injection
  Peak Plasma Concentration (Cmax)
Cochlear Perilymph Pharmacokinetics | within a 24 hour period after injection
  single time point measurement in each patient of drug in cochlear perilymph

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Eye and Ear Hospital, Melbourne, Victoria, Australia